CLINICAL TRIAL: NCT05077215
Title: A Phase 3, Randomized, Open-Label, Active-Controlled, Superiority Trial of EG007, Added to the Combination of Lenvatinib Plus Pembrolizumab vs. Lenvatinib Plus Pembrolizumab in Patients With Advanced Endometrial Cancer
Brief Title: Efficacy and Safety of a Repurposed Drug Added to the Combination of Len Plus Pem in Advanced Endometrial Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Evergreen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPC-EG-007-3.1
Record Dates: First submitted 2021-09-22; First posted 2021-10-14 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Advanced Endometrial Cancer
MeSH Terms: interventions — pembrolizumab; Injections; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: EG-007+ Len+Pem Regimen (Experimental)
  Interventions: Drug: EG-007; Drug: Pembrolizumab 100 mg/ 4 ml (25 mg/ml) Injection; Drug: Lenvatinib Capsules
- Arm 2: Len+Pem Regimen (Active Comparator)
  Interventions: Drug: Pembrolizumab 100 mg/ 4 ml (25 mg/ml) Injection; Drug: Lenvatinib Capsules

INTERVENTIONS:
Drug: EG-007 — A Repurposed Drug
  Arms: Arm 1: EG-007+ Len+Pem Regimen
Drug: Pembrolizumab 100 mg/ 4 ml (25 mg/ml) Injection — Pembrolizumab will be provided as a sterile, preservative-free, clear to slightly opalescent, colorless to slightly yellow solution that requires dilution for intravenous infusion. Each vial contains 100 mg of pembrolizumab in 4 mL of solution.
Drug: Lenvatinib Capsules — Lenvatinib will be provided as 4-mg and 10-mg capsules. Lenvatinib is formulated with calcium carbonate, mannitol, microcrystalline cellulose, hydroxypropylcellulose, low-substituted hydroxypropylcellulose, and talc.

SUMMARY:
This is a Phase 3, multicenter, randomized, open-label trial to evaluate whether EG-007 plus Len+Pem is superior to Len+Pem alone in patients with advanced endometrial cancer (Stage III or IV). This trial will be preceded by a safety lead-in study with up to 28 patients (the safety lead-in is a separate, free-standing protocol).

Approximately 450 patients will be randomized equally (1:1) to receive EG-007 plus Len+Pem or Len+Pem alone. The randomization will be stratified by the following stratification factors:

* Diagnosis Classification (advanced Stage III/IV vs. recurrent endometrial cancer)
* ECOG score at baseline (0 vs 1)
* Geographic region (Asia vs ROW)

ELIGIBILITY:
Inclusion Criteria:

1. Female, 18 years and older at the time of informed consent, who has a histologically confirmed diagnosis of endometrial carcinoma, endometroid histology, that is not MSI-H or dMMR.
2. Documented evidence of advanced (Stage III or IV), or recurrent EC.
3. Must have a recurrence or progressed on a platinum containing chemotherapy regimen and are not candidates for curative surgery or radiation
4. Has historical or fresh tumor biopsy specimen for confirmation of mismatch repair (MMR) status as not MSI-H or dMMR.
5. Has measurable or evaluable disease according to Response Evaluation Criteria In Solid Tumors (RECIST v1.1).
6. Is a candidate for initiation of treatment with the combined regimen of Keytruda plus Lenvima (Len+Pem) at the doses specified as the Len+Pem Regimen (per Labeling August 2021).
7. Life expectancy of 12 weeks or more.
8. Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 within 7 days of starting study treatment.
9. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP less than or equal to 150/90 mmHg at screening and no change in antihypertensive medications within 1 week prior to the first dose of study treatment.
10. Adequate renal function defined as creatinine less than or equal to 1.5 × ULN (upper limit of normal) or calculated creatinine clearance greater than or equal to 40 mL/min per the Cockcroft and Gault formula with creatinine levels greater than 1.5 × ULN.

Additional detail upon request.

Exclusion Criteria:

1. Brain metastasis: Brain metastases must be asymptomatic, fully treated and stable and not requiring steroids within 4 weeks prior to study treatment initiation.
2. Has carcinosarcoma (malignant mixed mullerian tumor), serous carcinoma, endometrial leiomyosarcoma and endometrial stromal sarcomas.
3. Has failed treatment of lenvatinib + pembrolizumab in prior lines of therapy.
4. Prior anticancer treatment within 28 days (or 5 times the half-life time, whichever is shorter) or any investigational agent within 30 days prior to the first dose of study drugs. All acute toxicities related to prior treatments must be resolved to Grade less than or equal to 1.
5. Participants must have recovered adequately from any toxicity and/or complications from major surgery prior to starting therapy.
6. Participants having greater than 1+ proteinuria on urinalysis will undergo 24-h urine collection for quantitative assessment of proteinuria. Participants with urine protein greater than or equal to 1 g/24-hour will be ineligible.
7. Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of the study drugs
8. Has a pre-existing greater than or equal (>=) Grade 3 gastrointestinal or non-gastrointestinal fistula.
9. Has radiographic evidence of major blood vessel invasion/infiltration.
10. Has clinically significant tumor bleeding within 2 weeks prior to the first dose of study treatment.

Additional detail upon request.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 35 Cycles of 21 days
  Progression-free survival (PFS) by RECIST v1.1 treatment vs. control group

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 35 Cycles of 21 days
  Objective Response Rate (ORR) treatment vs. control group
Overall survival (OS) | Up to 35 Cycles of 21 days
  Overall survival (OS) treatment vs. control group
Duration of response (DOR) | Up to 35 Cycles of 21 days
  Duration of response (DOR) treatment vs. control group
Disease control rate | Up to 35 Cycles of 21 days
  Disease control rate (DCR: CR + PR + stable disease [SD]) treatment vs. control group
Durable stable disease rate | Up to 35 Cycles of 21 days
  Durable stable disease rate (durable SD [SD ≥23 weeks]) treatment vs. control group
Clinical benefit rate | Up to 35 Cycles of 21 days
  Clinical benefit rate (CBR: CR, PR + durable SD) treatment vs. control group